CLINICAL TRIAL: NCT03930654
Title: Leveraging the Emergency Department to Engage African American Women in HIV Pre-Exposure Prophylaxis
Acronym: IWPrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mandy Hill, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-16-0892
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections
Keywords: African American women, HIV risk, substance use, sexual risk
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be assigned to either an intervention or usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPrEP Intervention (Experimental): iPrEP Intervention:
  * Women will receive the iPrEP intervention on an iPAD Air tablet device
  * iPrEP serves a dual role as a data collection instrument and an intervention--the survey incorporates brief, informational messages into a traditional survey instrument
  * iPrEP uses qualitative themes
  * iPrEP is divided into sections addressing factors with historical success at predicting pre-exposure prophylaxis (PrEP) adherence
  * Scales chosen to measure themes and sections were retained from the original HIV Prevention Trials Network (HPTN) 073 instrument
  * Scales were modified (in some cases) for cultural competency and tailoring to women
  Interventions: Behavioral: iPrEP; Behavioral: Usual Care
- Usual Care (Active Comparator): Control Intervention:
  * Women will receive usual care
  * Usual care includes an assessment visit with an emergency department (ED)-assigned social worker who specializes in substance use
  * Social worker will offer a list of substance abuse treatment referral agencies
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: iPrEP — * iPrEP transforms the standard emergency department (ED) visit experience through an intervention presented as a standard assessment that is equipped to: 1) increase knowledge of HIV transmission and 2) provide information on how to reduce an individual's risk for HIV.
  * Women will receive the iPrEP intervention on an iPAD Air tablet device
  * iPrEP serves a dual role as a data collection instrument and an intervention--the survey incorporates brief, informational messages into a traditional survey instrument
  * iPrEP uses qualitative themes
  * iPrEP is divided into sections addressing factors with historical success at predicting pre-exposure prophylaxis (PrEP) adherence
  * Scales chosen to measure themes and sections were retained from the original HIV Prevention Trials Network (HPTN) 073 instrument
  * Scales were modified (in some cases) for cultural competency and tailoring to women
  Arms: iPrEP Intervention
Behavioral: Usual Care — * Women will receive usual care
  * Usual care includes an assessment visit with an emergency department (ED)-assigned social worker who specializes in substance use
  * Social worker will offer a list of substance abuse treatment referral agencies

SUMMARY:
African American (AA) women are more vulnerable to HIV infection than other women. Truvada, when used as pre-exposure prophylaxis (PrEP), is one of the most effective approaches for HIV prevention; however, PrEP use among AA women remains low and has not responded to traditional interventions. This study proposes for the first time an innovative computer-based motivational intervention, increasing PrEP uptake (iPrEP), which couples motivational messages woven into a traditional survey to raise awareness of risky sex and substance use behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Current HIV negative status (based on ED' HIV test outcome)
* Condomless sex in the last 3 months
* Substance use in the last 3 months
* HIV testing during ED visit (usual care)
* Has a non-emergent health condition
* Has a working mobile device with them

Exclusion Criteria:

* Ineligible for PrEP (see eligibility criteria to the right)
* Assigned male at birth
* An HIV positive status
* Currently taking medication that are known contraindications for PrEP (brand name: Truvada)
* Currently on PrEP

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who were assigned a male sex at birth are excluded from study participation.
Enrollment: 40 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with an increased willingness for pre-exposure prophylaxis (PrEP) uptake | 1 month
  Participants will be assessed for social norms and risk.
Number of participants with an increased willingness for pre-exposure prophylaxis (PrEP) uptake | 3 months
  Participants will be assessed for social norms and risk.
Number of participants with an increased willingness for pre-exposure prophylaxis (PrEP) uptake | 6 months
  Participants will be assessed for social norms and risk.

SECONDARY OUTCOMES:
Number of participants with decreased high risk sex | 1 month
Number of participants with decreased high risk sex | 3 months
Number of participants with decreased high risk sex | 6 months
Number of participants with decrease in substance use | 1 month
Number of participants with decrease in substance use | 3 months
Number of participants with decrease in substance use | 6 months
Number of participants with a new sexually transmitted disease diagnosis | 1 month
Number of participants with a new sexually transmitted disease diagnosis | 3 months
Number of participants with a new sexually transmitted disease diagnosis | 6 months
Number of participants with HIV seroconversion | 1 month
Number of participants with HIV seroconversion | 3 months
Number of participants with HIV seroconversion | 6 months
iPrEP feasibility and acceptability as assessed by the number of participants who believe that they had more information to make a better decision about being in a PrEP program after completing the survey intervention | baseline
  As part of the survey, participants will be asked if they believe that they had more information to make a better decision about being in a PrEP program after completing the survey intervention.
iPrEP feasibility and acceptability as assessed by how much participant liked or disliked completing the survey | baseline
  As part of the survey, participants will asked "How much did you like or dislike completing this questionnaire?" and will choose one of the following 5 categorical choices: Liked it, Liked it somewhat, Neither liked nor disliked it, Disliked it somewhat, Disliked it
iPrEP feasibility and acceptability as assessed by how often participants relied on the survey questions being read aloud to be able to answer them | baseline
  As part of the survey, participants will asked "As you completed this questionnaire, how often did you rely on the questions being read aloud to be able to answer them?" and will choose one of the following 4 categorical choices: For all the questions, For most of the questions, For some of the questions, For none of the questions
iPrEP feasibility and acceptability as assessed by number of participants who needed help from site staff in order to complete the survey | baseline
  As part of the survey, participants will be asked if they needed help from site staff in order to complete the survey.
iPrEP feasibility and acceptability as assessed by the kind of help that participants needed from site staff in order to complete the survey | baseline
  As part of the survey, participants will asked "What kind of help did you need? Please check all that apply" and will choose among the following categorical 4 choices: I had to have some of the questions explained to me, I needed help using the iPAD, I needed to have the questionnaire read to me by a staff member, I needed help for a different reason
iPrEP feasibility and acceptability as assessed by how participants felt about the length of the survey | baseline
  As part of the survey, participants will asked how they felt about the length of the survey and will choose one of the following 3 categorical choices: Too long, Too short, The right length

CONTACTS AND LOCATIONS:
Overall Officials: Mandy J Hill, DrPH, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hill MJ, Heads AM, Suchting R, Stotts AL. A survey with interventional components delivered on tablet devices versus usual care to increase pre-exposure prophylaxis uptake among cisgender Black women: a pilot randomized controlled trial. BMC Infect Dis. 2023 Jan 27;23(1):57. doi: 10.1186/s12879-023-08019-z. PMID 36707778